CLINICAL TRIAL: NCT02382263
Title: Phase I/II Study to Assess the Efficacy and Safety of Nab-paclitaxel in Combination With Gemcitabine for the Treatment of Fragile Patients With Advanced or Metastatic Pancreatic Cancer
Brief Title: Nab-paclitaxel in Combination With Gemcitabine in Fragile Patients With Advanced Pancreatic Cancer
Acronym: FRAGANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PH Research, S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHR-2012-01
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Advanced pancreatic cancer; Fragile; Nab-paclitaxel
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm B (Experimental): Nab-paclitaxel 150 mg/m2 + Gemcitabine 1000 weeks 1,3/4
  Interventions: Drug: Nab-paclitaxel 150 mg/m2 + Gemcitabine 1000 weeks 1,3/4
- Arm C (Experimental): Nab-paclitaxel 100 mg/m2 + Gemcitabine 1000 weeks 1,2,3/4
  Interventions: Drug: Nab-paclitaxel 100 mg/m2 + Gemcitabine 1000 weeks 1,2,3/4
- Arm D (Experimental): Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 weeks 1,3/4
  Interventions: Drug: Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 weeks 1,3/4
- Arm E (Experimental): Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 weeks 1,2,3/4
  Interventions: Drug: Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 weeks 1,2,3/4

INTERVENTIONS:
Drug: Nab-paclitaxel 150 mg/m2 + Gemcitabine 1000 weeks 1,3/4 — Nab-paclitaxel 150 mg/m2 + Gemcitabine 1000 days 1 & 15 in a 28 days cycle
  Arms: Arm B
Drug: Nab-paclitaxel 100 mg/m2 + Gemcitabine 1000 weeks 1,2,3/4 — Nab-paclitaxel 100 mg/m2 + Gemcitabine 1000 days 1,8 & 15 in a 28 days cycle
  Arms: Arm C
Drug: Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 weeks 1,3/4 — Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 days 1 & 15 in a 28 days cycle
  Arms: Arm D
Drug: Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 weeks 1,2,3/4 — Nab-paclitaxel 125 mg/m2 + Gemcitabine 1000 days 1,8 & 15 in a 28 days cycle
  Arms: Arm E

SUMMARY:
In the list of cancer mortality by type of cancer pancreatic cancer ranks 4th in USA and the 6th in Europe. The estimated figures for 2010 in the USA were 42,000 new cases and 36,000 deaths from pancreatic cancer. The survival rate at 5 years after diagnosis is 4.6% in the USA. In Europe the figures are similar, with survival at 1, 3 and 5 years of 16%, 6% and 4%, respectively. Most patients are diagnosed in advanced stages that are no longer operable, so that treatment goals are often the prolongation of survival and palliation of symptoms.

The aim of the study is to explore whether the new combination nab-paclitaxel plus gemcitabine is a therapeutic advance for this fragile population for which it is assumed that some modifications in dose and schedule of administration may be necessary in patients with good performance status. It is ultimately to find out the clinical benefit of this combination, but first making sure that dose and schedule of the combination are tolerable for these fragile patients.

For this, the investigators have chosen a design that includes two stages: the first step aimed at choosing the safest treatment regimen for these patients among a group of treatment regimens used in other clinical trials. The second step will evaluate the effectiveness of the two regimens with the better results in the previous step.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older;
* Patients with histological or, if not possible, cytologic confirmed adenocarcinoma of the pancreas.
* Patients with metastatic pancreatic cancer;
* Patient with an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) = 2
* Adequate hematopoietic, hepatic and renal function:
* Neutrophil count >= 1.5 x 10*9/L;
* Platelet count >= 100 x 10*9/L;
* Bilirubin <= 1.5 x ULN;
* AST and/or ALT <= 2.5 x ULN;
* Serum creatinine <= 1.5 x ULN.
* Investigators must ensure that patients enrolled in the study will be available for all study procedures, including tumor biopsy, chemotherapy treatment, and follow up.
* Investigators must ensure that patients have the ability to understand the requirements of the study and provide signed informed consent.
* Women of childbearing potential and men who wish to participate in the study must agree to use adequate contraception since the signing of informed consent until at least 3 months after stopping the study medication;
* Signed Informed Consent.

Exclusion Criteria:

* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with patient eligibility for treatment;
* History of any psychiatric condition that might impair patient?s ability to understand or to comply with the requirements of the study or to provide informed consent;
* Concurrent anticancer therapy;
* Pregnant or breast-feeding women (documented methods of birth control are required in those with reproductive potential);
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs;
* History of life threatening reaction to gemcitabine or abraxane;
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) <=1.
* Previous treatment with chemotherapy or chemoradiotherapy for advanced pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
PHASE I: To select the schemes with the best therapeutic indexes of the combination of gemcitabine and nab-paclitaxel in fragile patients with advanced pancreatic cancer. | Up to 2 months
  Phase I: Therapeutic index. Criteria: Early mortality all causes at 30 and 60 days, Adverse Events grade 3 and 4, treatment discontinuation due to toxicity and relative dose intensity
PHASE II: Evaluate the effectiveness of two selected schemes of gemcitabine and nab-paclitaxel, vs. gemcitabine alone. (Six months overall survival) | Up to 6 months
  Six months overall survival

SECONDARY OUTCOMES:
Phase I: evaluate safety profile of gemcitabine and nab-paclitaxel schemes. (Number of events per patient according to NCI-CTC-AE criteria) | Up to 6 months
  Number of events per patient according to NCI-CTC-AE criteria
Phase I: evaluate objective response rate. (Response rate will be evaluated according RECIST criteria) | Up to 6 months
  Response rate will be evaluated according RECIST criteria
Phase II: progression free survival (Time from randomization to disease progression according RECIST criteria) | Up to 8 months
  Time from randomization to disease progression according RECIST criteria
Phase II: objective response rate (Response rate will be evaluated according RECIST criteria) | Up to 6 months
  Response rate will be evaluated according RECIST criteria
Phase II: to explore changes induced by treatment on tumor Marker CA19.9 | Up to 8 months
Phase II: change in FAP and Cav-1 tumor markers as an inidicatior of treatment efficacy | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, Study Chair — Hospital Universitario Madrid Sanchinarro; Fernando Rivera, MD, Principal Investigator — HOSPITAL UNIVERSITARIO MARQUÉS DE VELDECILLA; Teresa Macarulla, MD, Principal Investigator — Hospital Vall d'Hebron; Carmen Guillén, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Rafael López, MD, Principal Investigator — COMPLEXO HOSPITALARIO UNIVERSITARIO DE SANTIAGO; Roberto Pazo, MD, Principal Investigator — Hospital Miguel Servet; Manuel Valladares, MD, Principal Investigator — COMPLEXO HOSPITALARIO UNIVERSITARIO A CORUÑA; Roberto P Díaz, MD, Principal Investigator — Hospital Universitario La Fe; Inmaculada Alés, MD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL DE MÁLAGA; Joaquina Martínez, MD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL VIRGEN DE LAS NIEVES; Adelaida La Casta, MD, Principal Investigator — Hospital Donostia; Rut Vera, MD, Principal Investigator — Complejo Hospitalario de Navarra; Andrés Muñoz, MD, Principal Investigator — COMPLEJO HOSPITALARIO GREGORIO MARAÑÓN; José I Martín, MD, Principal Investigator — HOSPITAL UNIVERSITARIO FUNDACIÓN JIMÉNEZ DIAZ; Javier Sastre, MD, Principal Investigator — Hospital San Carlos, Madrid
Locations (15):
- Spain (15):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Cosuña
  - Hospital Universitari Vall D'Hebron, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Complejo Hospitalario Regional Virgen de Las Nieves, Granada, Granada
  - Complejo Hospitalario Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón Y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid, Madrid
  - Complejo Hospitalario Regional de Málaga, Málaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitari I Politècnic La Fe, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza